CLINICAL TRIAL: NCT05653765
Title: Prognostic Value of the Angio-based Microvascular Resistance Use One Single Angiographic View Measured After Primary Percutaneous Coronary Intervention in ST-segment Elevation Myocardial Infarction Patients
Brief Title: Prognostic Value of the AMR Measured After PPCI in STEMI Patients
Acronym: EARLYMYOAMR
Status: Active, not recruiting | Type: Observational
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Other Study IDs: HenanICE202201
Record Dates: First submitted 2022-11-04; First posted 2022-12-16 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Coronary Heart Disease; ST Elevation Myocardial Infarction
MeSH Terms: conditions — Coronary Disease; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- diagnostic cohort/derivation cohort: The diagnostic/derivation cohort included STEMI patients who underwent PCI within 12 hours and CMR. The optimal AMR cutoff value for diagnosing CMD using CMR was determined by analyzing ROC curves.
- prognostic cohort/validation cohort: The prognostic cohort enrolled STEMI patients who underwent PPCI within 12 hours. All patients were followed up for at least 1 year.

SUMMARY:
The goal of this observational study is to learn about in STEMI with Primary PCI Patients. The main questions it aims to answer are:

* To determine the value of AMR in predicting the long-term clinical prognosis of patients with STEMI after PPCI, and to find the best cut-off value.
* Analyze the factors of PPCI affecting AMR and explore the effective measures of PPCI microcirculation protection.

Radiographic images of STEMI receiving primary PCI treatment in several chest pain centers in China will be included. The last image of the infarct-related vessel will be used as a target to calculate its AMR. The relationship between AMR and long-term clinical prognosis was analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or older
* Type 1 myocardial infarction
* Receive PPCI

Exclusion Criteria:

* Failed to identify culprit vessels.
* Structural heart disease with moderate to severe aortic valve or mitral regurgitation and or stenosis that may affect cardiac function
* Dialysis patients with severe renal insufficiency
* Severe and uncontrollable arrhythmia
* Complicated with dilated cardiomyopathy
* Unable to tolerate dual antiplatelet therapy
* Severe and uncontrollable anemia
* Hyperthyroidism
* TIMI blood flow 0-1 grade after PPCI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent PPCI due to STEMI in several chest pain centers in China from January 1, 2012 to October 1, 2022
Sampling Method: Non-Probability Sample
Enrollment: 2663 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
MACEs | 12 months
  cardiac death, hospitalization for heart failure, target vessel revascularization，non-fatal MI

SECONDARY OUTCOMES:
cardiac death | 12 months
  All cause deaths will be considered cardiac unless a definite noncardiac cause can be established.
hospitalization for heart failure | 12 months
  Hospitalization for heart failure was defined as admission because of new or deteriorating signs and symptoms of heart failure combined with the findings of noninvasive imaging or elevated B-type natriuretic peptide(BNP) and/or N-terminal pro-BNP concentration, and a discharge diagnosis of congestive heart failure.
target lesion revascularization | 12 months
  The following 3 conditions need to be met at the same time:
  1. The new stenosis that developed within previously treated coronary segments and within 5 mm of their borders;
  2. The new stenosis resulted in the vessel μQFR ≤ 0.80;
  3. The patient subsequently underwent repeat PCI or coronary artery bypass grafting (CABG).
Repeated myocardial infarction | 12 months
  Repeated myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Muwei Li, MD, Study Chair — Fuwai central China cardiovascular hospotial
Locations (5):
- China (5):
  - Shangqiu first people's Hospital, Shangqiu, Henan
  - Department of Cardiology, First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Yongcheng Central Hospital, Yongcheng, Henan
  - Fuwai central China cardiovascular Hospital, Zhengzhou, Henan
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University,, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No
The personal information of a large number of patients is involved. IPD is not provided to protect the privacy of participants.